CLINICAL TRIAL: NCT01350024
Title: Comparison of Postoperative Pain With Two Different Types of Local Anesthesia in Surgery for a Drooping Eyelid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Dr. Wendy Lee, Assoc. Professor of Clinical, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20100631
Record Dates: First submitted 2011-05-05; First posted 2011-05-09 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Blepharoptosis
Keywords: Conjunctival Mullerectomy; Blepharoptosis; Ptosis surgery; Pain Control
MeSH Terms: conditions — Blepharoptosis; Agnosia | interventions — Lidocaine; Indicator Dilution Techniques; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Frontal Nerve Block (Active Comparator): Patients will receive a frontal nerve block for anesthesia
  Interventions: Procedure: Frontal nerve block with 2% lidocaine with 1:100,000 dilution of epinephrine
- Subconjucntival Injection (Active Comparator): Patients will receive a subconjunctival injection for anesthesia
  Interventions: Procedure: Subconjunctival injection of 2% lidocaine with 1:100,000 dilution with epinephrine

INTERVENTIONS:
Procedure: Frontal nerve block with 2% lidocaine with 1:100,000 dilution of epinephrine — Frontal Nerve Block 5 cc will be administered preoperatively once.
  Arms: Frontal Nerve Block
Procedure: Subconjunctival injection of 2% lidocaine with 1:100,000 dilution with epinephrine — Patients will receive a 1.5 cc dose of subconjunctival lidocaine as above
  Arms: Subconjucntival Injection

SUMMARY:
Conjunctival Mullerectomy is a well known procedure used to correct upper lid ptosis via a posterior approach. Patients who undergo this procedure are often given local anesthesia to alleviate intraoperative and postoperative pain. Local anesthesia can be given via frontal nerve block or subconjunctival injection combined with sedation in most cases. Both techniques are currently acceptable options for local anesthesia, however postoperative pain has not been systematically evaluated between these two techniques.

The investigators aim to compare intra-operative and postoperative pain with these two techniques in patients undergoing conjunctival Mullerectomy for ptosis repair. Patients will be randomized to receive local anesthesia via frontal nerve block or via subconjunctival injection. In addition, the investigators will measure the surgical outcomes of the ptosis surgery with standard measures.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Patient with ptosis that requires correction
* Patient is able to consent for themselves

Exclusion Criteria:

* Patient unable to complete survey
* Patient had prior lid surgery
* Patient taking chronic pain medication

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-05-01 (Actual); Primary Completion 2016-07-30 (Actual); Study Completion 2016-07-30 (Actual)

PRIMARY OUTCOMES:
Pain control | 24 hour after surgery
  Patients will be asked to complete a survey regardning pain assessment twenty-four hours after completion of surgery.

SECONDARY OUTCOMES:
Efficacy of ptosis surgery | 2 months
  Standard measures include marginal reflex distanced, palpebral fissure and levator fucntion will be used to assess the efficacy of the ptosis surgery and compared to the type of anesthesia the patient was given.
Pain Control | 1 hour after surgery
  completion of survey to assess pain after surgery has been completed.

CONTACTS AND LOCATIONS:
Locations (1):
- Bascom Palmer Eye Institute, Miami, Florida, United States